CLINICAL TRIAL: NCT04714450
Title: Assessing the Efficacy and Repeatability of the Mannheim Multicomponent Stress Test
Brief Title: Assessing the Repeatability of a Psychological Stress Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Collaborators: Danone Nutricia Research (Industry)
Responsible Party: Principal Investigator, Daniel Kashi, Doctor, Liverpool John Moores University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ORION Study 1A
Record Dates: First submitted 2021-01-12; First posted 2021-01-19 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Stress, Physiological; Stress, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: The investigators propose a parallel experimental trial examining physiological and psychological responses to a socio-evaluative stress task (The Mannheim Multicomponent Stress Test; MMST) under laboratory conditions. Participants will be tested on three occasions in a randomised order, with each trial separated by 7 days. On two occasions, participants will be complete a socially evaluated math-based serial addition task whilst simultaneously viewing a series of positive and negative images and in the presence of white noise (duration ~ 5 minutes). On the other occasion, participants will rest quietly and will be exposed to a short film and some images that are not designed to induce anxiety or stress for the same duration as the stress test in the stress induction room. The non-stress control condition, will occur either 1-week preceding or 1-week following both MMST trials, thereby controlling for order effects influencing baseline physiological and psychological outcome measures.
Who Masked: Outcomes Assessor
Masking Description: Saliva samples will be identified by participant identification number only. Technicians assessing levels of biological measures in these samples will be blind to condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MMST control (No Intervention)
- MMST+ (Experimental)
  Interventions: Behavioral: Experimental: MMST+

INTERVENTIONS:
Behavioral: Experimental: MMST+ — The format of the MMST will remain the same; however, the white noise, images and math task will be modified to mitigate habituation effects.
  Arms: MMST+

SUMMARY:
To establish the efficacy and repeatability of a suitable psychological stress test. The Mannheim Multicomponent Stress Test (MMST) is a validated laboratory stress test that combines cognitive, emotional, acoustic and motivational stress components. Despite the test increasing self-reported levels of stress, meaningful changes in saliva cortisol are typically observed in only half of all participants. In addition, the MMST is susceptible to habituation of the cortisol response upon repeated exposures, limiting its current usefulness for repeated measures. Given the multicomponent nature of the MMST, there is potential for components of the test to be manipulated to overcome these limitations i.e., increase the magnitude of the saliva cortisol response and mitigate against habituation effects. In addition, a supplementary topic of interest is to what extent cortisol responses to acute laboratory stress tests, like the MMST, relate to the well described rise in morning cortisol ~30 minutes after awakening. This may be of clinical relevance given that blunted cortisol response upon awakening and in response to acute psychological stress tests have been associated with poor health outcomes.

The primary objective of the current study is to investigate if the MMST elicits a meaningful increase in saliva cortisol.

The secondary objective is to investigate the efficacy of mitigation strategies to overcome habituation to the MMST.

A supplementary objective is to to investigate the relationship between the saliva cortisol response upon awakening and the saliva cortisol response to the MMST.

ELIGIBILITY:
Inclusion Criteria:

Participants who…

* have read and signed the study informed consent
* are healthy, recreationally active men and women aged 18-35 years
* test negative for coronavirus (COVID-19)
* are willing to provide saliva samples throughout and complete the MMST through the duration of the study
* are using monophasic birth control (women only)

Exclusion Criteria:

Participants who…

* have a recent history or are a current smoker
* are currently taking prescription/Over-the-counter medication
* consume ≥ 91 units of alcohol per month
* have a clinically diagnosed history of cardiovascular and/or metabolic disease including diabetes and abnormal blood pressure
* are pregnant
* have a recent or ongoing viral or bacterial illness in past 4 weeks
* test positive for coronavirus (COVID-19)
* have a clinically diagnosed psychiatric disorder
* have a clinically diagnosed sleeping disorder
* have a clinically diagnosed gambling addiction
* BMI ≥ 30 kg/m2 - calculated in the online health screening questionnaire
* report unusually high levels of recent or ongoing life stress over the last month; as assessed by the perceived stress scale (PSS) i.e. rating ≥ 13 indicates high perception of recent and ongoing life stress
* Endurance trained or engage in ≥3.5 hours of physical activity a week

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Change in saliva cortisol (pre-post MMST) | Change from 5 minutes pre to peak post stress test/no stress control condition
  Changes in the concentration of saliva free cortisol assessed by ELISA.
Change in subjective stress response (Subjective stress scale) (0-9 Likert scale) | Change from 5 minutes pre to immediately post stress test/no stress control condition
  Questionnaire comprised of a 10-point rating scale from 0 to 9 (0 - no subjective stress experience at all; 9 - extreme experience of subjective stress experience.
Heart rate | Continuously assessed from 30 minutes before to 60 minutes after the stress tests and control tests
  Continuous measurement of heart rate will be assessed using a telemetric chest strap.

SECONDARY OUTCOMES:
Change in emotional response to stress | Change from 5 minutes pre to immediately post stress test/no stress control condition
  Questionnaire used to determine the extent to which participants felt the MMST was difficult, challenging, and upsetting. Using a 7-pt scale (1 = not at all; 7 = extremely) participants rate their level of nervousness during the laboratory task. Participants will also rate the level of effort they put into the task on a scale ranging from 1 (didn't try at all) to 7 (tried as hard as I could), which will be used as a manipulation check.
Rumination measure | Assessed +60 minutes after the stress tests and no stress control condition
  Questionnaire used to determine the extent of rumination about an induced stressful situation. Using a 7-pt scale (1= not at all, 7 = all the time), participants indicate the extent to which they; thought about the test (stress test and control) after having completed it, criticised themselves about not performing well, thought about other past experiences of being evaluated, thought about the anxiety they felt during the task.

OTHER OUTCOMES:
Saliva cortisol awakening response (CAR) | Assessing upon awakening, and every 15 minutes for the first 45 minutes after awakening (i.e. +15, +30, +45, +60 minutes after awakening)
  A biomarker for Hypothalamic Pituitary Adrenal activity; a naturally occurring increase in cortisol upon waking, assessed by ELISA.
Salivary alpha amylase (sAA) | Change from 5 minutes pre to immediately post stress test/no stress control condition
  a biomarker for stress-induced activity of the sympathetic nervous system (SNS), assessed by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Neil P Walsh, PHD, Principal Investigator — Liverpool John Moores University
Locations (1):
- Faculty of Science, Liverpool John Moores University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No